CLINICAL TRIAL: NCT05146505
Title: Analysis of Circulating miRNAs as Potential Biomarkers of Diagnosis and Prognosis in High Grade Serous Ovarian Cancer
Brief Title: miRNAs in High Grade Serous Ovarian Cancer
Acronym: MIROC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Anna Myriam Perrone, MD, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: 788/2021/Sper/AOUBo
Record Dates: First submitted 2021-11-20; First posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: High Grade Serous Ovarian Cancer
Keywords: miRNAs

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — RNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
High grade serous ovarian cancer represents the gynecological malignancy with the highest incidence of mortality. Decision-making tools are currently limited to the use of standard imaging modalities and analysis of serum biomarkers, such as CA 125, which often have low specificity and sensitivity. Recently, a growing research interest has been aimed at so-called circulating microRNAs (miRNAs). Indeed, it has been observed that miRNAs are abundantly present in all biological fluids and play the key role of messengers in intercellular communication. Cancer cells have a rapid turnover which results in a continuous release of nucleic acids and vesicles derived from the tumor itself, such as the tumor cells themselves that separate from the tumor mass to enter the bloodstream. Given their important role as modulators of gene expression, in order to preserve their integrity, miRNAs are encapsulated in specific vesicles, in order to prevent their degradation by the enzymes present in biological fluids. In this context, the chance of monitoring the expression levels of specific miRNAs represents a very interesting option both for an early diagnosis and for monitoring the clinical response to pharmacological treatment. Currently, there are no non-invasive approaches to monitor the clinical outcome in real time, while the identification of circulating biomarkers would allow prompt intervention, possibly modifying the pharmacological management in case of progression.

ELIGIBILITY:
Inclusion Criteria:

* age>18
* Histological diagnosis of epithelial ovarian cancer
* Patients eligible for surgery
* Patients followed in the clinical care pathway c / o oncological gynecology (surgery and follow up)
* informed consent

Exclusion Criteria:

* Patients with HCV, HBV and HIV
* Patients with other malignancies diagnosed less than 5 years prior to the diagnosis of ovarian malignancy
* Ovarian metastases of primary neoplasms of other organs
* Presence of ascites for non-neoplastic causes

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women with high grade serous ovarian cancer
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Longitudinal miRNAs analysis over chemotherapy | 2 years
  Evaluation of miRNA expression in longitudinal blood samples collected during every follow-up

SECONDARY OUTCOMES:
Associaition miRNA-clinico-pathological data | 2 years
  Correlation between miRNAs deregulation and clinico-pathological and molecular data

CONTACTS AND LOCATIONS:
Overall Officials: Anna Myriam Perrone, Principal Investigator — IRCCS Azienda Ospedaliera-Universitaria di Bologna
Locations (1):
- IRCCS- Azienda Ospedaliera-Universitaria di Bologna, Bologna, Bo, Italy

IPD SHARING:
Plan to Share IPD: No